CLINICAL TRIAL: NCT05841654
Title: Effect of Azilsartan on the Incidence of Atrial Fibrillation in Patients With Hypertension Combined With Left Ventricular Hypertrophy
Brief Title: Effect of Azilsartan on Atrial Fibrillation in Patients With Hypertension
Acronym: AZAF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022-CCA-HX-009
Record Dates: First submitted 2023-03-23; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hypertension; Atrial Fibrillation
Keywords: Azilsartan; Atrial Fibrillation; Hypertension; Left Ventricular Hypertrophy
MeSH Terms: conditions — Hypertension; Atrial Fibrillation; Hypertrophy, Left Ventricular | interventions — azilsartan

STUDY DESIGN:
Intervention Model Description: In the study, the selected patients would be randomly divided into the Azilsartan treatment group and the conventional treatment group, and all the selected patients would be regularly followed up for 12 months. In the Azilsartan group, Azilsartan will be added in or switched to the original antihypertensive treatment plan, starting as 20 mg Qd, and gradually increased to 40 mg Qd according to the blood pressure. If the blood pressure is still not be controlled, antihypertensive drugs other than angiotensin-converting enzyme inhibitor (ACEI), ARB or angiotensin receptor blocker and neprilysin inhibitor (ARNI) will be added until the blood pressure is controlled. In the routine treatment group, antihypertensive treatment programs other than ACEI, ARB or ARNI will be adopted, and the use of antihypertensive drugs will be adjusted until the blood pressure control is controlled.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azilsartan treatment group (Experimental): In the Azilsartan group, Azilsartan will be added in or switched to the original antihypertensive treatment plan, starting as 20 mg Qd, and gradually increased to 40 mg Qd according to the blood pressure. If the blood pressure is still not be controlled, antihypertensive drugs other than ACEI, ARB or ARNI will be added until the blood pressure is controlled.
  Interventions: Drug: Azilsartan or antihypertensive drugs other than ACEI, ARB or ARNI
- Conventional treatment group (Active Comparator): In the routine treatment group, antihypertensive treatment programs other than ACEI, ARB or ARNI will be adopted, and the use of antihypertensive drugs will be adjusted until the blood pressure control is controlled.
  Interventions: Drug: Azilsartan or antihypertensive drugs other than ACEI, ARB or ARNI

INTERVENTIONS:
Drug: Azilsartan or antihypertensive drugs other than ACEI, ARB or ARNI — The patient's ECG information will be monitored through the ECG monitoring patch, and the time of the first atrial fibrillation event will be recorded. Monitoring whether the patient's blood pressure is controlled dynamically, using echocardiography to evaluate cardiac function, and using scales to assess the quality of life.

SUMMARY:
Hypertension and atrial fibrillation (AF) are two major public health problems worldwide. Hypertension is an important risk factor for AF, and the combination of which could significantly increase the risk of cardiovascular adverse events, and result greater disability rate and mortality.

Hypertension can stimulate cardiomyocytes apoptosis, drive renin-angiotensin-aldosterone system (RAAS) activation, lead to left ventricular hypertrophy (LVH) and finally result in the structure remodeling of the atrium, which can trigger AF development through influence on myocardial electrical activity. Previous studies have found that angiotensin receptor blockers (ARB) seem to be more efficient in preventing AF when hypertension combined heart failure or LVH, but not completely clear in others with hypertension.

Azilsartan is a new ARB, it replaces the tetrazole ring of the traditional ARB with the oxadiazole ring, which making it binds to the angiotensin type 1 (AT1) receptor more tightly, dissociate more slowly, and has a stronger antihypertensive effect. It was reported that Azilsartan could inhibit cell proliferation, reduce inflammation and oxidative stress. However, whether Azilsartan can reduce the risk of AF in hypertensive patients, and the possible corresponding mechanism is still unclear.

Accordingly, the investigators designed this study intending to evaluate the effect of Azilsartan on the incidence of AF in hypertensive patients combined with LVH, and to explore the possible mechanism. This study is a practical, multicenter randomized controlled research method, the investigators will include 400 patients with hypertension and LVH who meet the inclusion criteria in Beijing Tsinghua Changgung Hospital and other centers. The patients would be divided into the Azilsartan group and conventional treatment group randomly, and be followed up regularly for 12 months. The incidence of AF in the two groups would be compared through the flexible intelligent ECG monitoring system, and the optimal blood pressure control, also the left ventricular hypertrophy and left atrial function would be evaluated.

This study will provide evidence for the use of Azilsartan in blood pressure control and lower risk for AF patients with hypertension and LVH. It will be benefit for improving prognosis of patients with hypertension combined LVH, reducing the incidence of AF, and achieving good social economic effects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Satisfied the diagnostic criteria for hypertension in the 2020 International Society of Hypertension Global Practice Guidelines for Hypertension.
* Blood pressure control fails to meet one of the following conditions: office blood pressure ≥ 140/90mmHg; ambulatory blood pressure monitoring daytime average blood pressure ≥ 135/85mmHg or nighttime average blood pressure ≥ 120/70mmHg; home monitoring blood pressure ≥ 135/85mmHg.
* Echocardiography shows that the left ventricular wall thickness is ≥11 mm, or the left ventricular mass index (LVMI) is >95 g/m2 (female), 115 g/m2 (male).

Exclusion Criteria:

* Secondary hypertension.
* Confirmed diagnosis of persistent atrial fibrillation.
* Severe liver and kidney disease (eGFR<30 mL/min/1.73m2), severe lung disease, malignant tumor and mental illness history.
* Pregnant women, women of childbearing age who plan to become pregnant during the study or who cannot use effective contraception during the study
* Illness leading to life expectancy <12 months.
* Not signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and burden of atrial fibrillation | The patient's ECG information will be recorded once a month, and be continuously monitored for 7 days at each time. A 24-hour Holter electrocardiogram was performed within 48 weeks.
  In this study, atrial fibrillation includes both paroxysmal or persistent atrial fibrillation. Paroxysmal atrial fibrillation refers to that lasts for more than 30 seconds but less than 7 days, and the persistent one refers to that lasts over 7 days. Atrial fibrillation burden is defined as the percentage of analyzable wear time in AF.

SECONDARY OUTCOMES:
Control of Blood pressure | Patients will conduct self-test blood pressure 3 days a week, once in the morning and once in the evening. A 12-week interval is used to calculate the TITRE values of the two groups of patients at 0-12 weeks, 13-24 weeks, 25-36 weeks, and 37-48 weeks.
  In this study, the percentage time to achieve blood pressure target (TITRE) and ambulatory blood pressure monitoring will be used to evaluate the achievement of blood pressure target. Greater percentage time at target (TITRE) was associated with lower risk of incident cardiovascular diseases and was an effective predictor of clinical outcomes, with a high clinical relevance and actionability. The standard calculation method of TITRE is based on that reported in previous studies.
Evaluation of left ventricular hypertrophy and left atrial dimension | From baseline to the end of study.
  Two-dimensional transthoracic echocardiography (2DE) diastolic interventricular septal thickness (IVST) or left ventricular posterior wall thickness (PWT) and left ventricular mass index (LVMI) will be used to evaluate left ventricular hypertrophy. According to the guidelines, IVST or PWT ≥ 11mm, LVMI > 95g/m2 (female)/115 g/m2 (male) is defined as left ventricular hypertrophy. Left atrial dimension is evaluated by left atrial volume index (LAVI). Left atrial volume is measured by two-dimensional echocardiography, and the left atrial volume index (LAVI) is obtained by correcting body surface area.
Healthy quality of life | From baseline to end of study
  In this study, three-level EuroQol five-dimensions (EQ-5D-3L) will be used to assess the patient's quality of life, and the difference in the change in the quality of life between the two groups will be compared. The EQ-5D-3L is a self-assessment scale which includes five dimensions: mobility, self-care, daily activities, pain or discomfort, and depression. There are three categories of options for each dimension (Normal, Moderately Restricted, Severely Restricted). This commonly used health utility measure converts quality of life and health status into quality-adjusted life years (QALYs).

CONTACTS AND LOCATIONS:
Overall Officials: He Rong, M.D., Ph.D, Study Chair — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Benjamin EJ, Muntner P, Alonso A, Bittencourt MS, Callaway CW, Carson AP, Chamberlain AM, Chang AR, Cheng S, Das SR, Delling FN, Djousse L, Elkind MSV, Ferguson JF, Fornage M, Jordan LC, Khan SS, Kissela BM, Knutson KL, Kwan TW, Lackland DT, Lewis TT, Lichtman JH, Longenecker CT, Loop MS, Lutsey PL, Martin SS, Matsushita K, Moran AE, Mussolino ME, O'Flaherty M, Pandey A, Perak AM, Rosamond WD, Roth GA, Sampson UKA, Satou GM, Schroeder EB, Shah SH, Spartano NL, Stokes A, Tirschwell DL, Tsao CW, Turakhia MP, VanWagner LB, Wilkins JT, Wong SS, Virani SS; American Heart Association Council on Epidemiology and Prevention Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2019 Update: A Report From the American Heart Association. Circulation. 2019 Mar 5;139(10):e56-e528. doi: 10.1161/CIR.0000000000000659. No abstract available. PMID 30700139
- [Background] Zhou Z, Hu D. An epidemiological study on the prevalence of atrial fibrillation in the Chinese population of mainland China. J Epidemiol. 2008;18(5):209-16. doi: 10.2188/jea.je2008021. Epub 2008 Sep 8. PMID 18776706
- [Background] Encephalopathy from hyponatremia. Ann Intern Med. 1990 Jul 1;113(1):84-6. doi: 10.7326/0003-4819-113-1-84_3. No abstract available. PMID 2350117
- [Background] Gumprecht J, Domek M, Lip GYH, Shantsila A. Invited review: hypertension and atrial fibrillation: epidemiology, pathophysiology, and implications for management. J Hum Hypertens. 2019 Dec;33(12):824-836. doi: 10.1038/s41371-019-0279-7. Epub 2019 Nov 5. PMID 31690818
- [Background] Chung SC, Pujades-Rodriguez M, Duyx B, Denaxas SC, Pasea L, Hingorani A, Timmis A, Williams B, Hemingway H. Time spent at blood pressure target and the risk of death and cardiovascular diseases. PLoS One. 2018 Sep 5;13(9):e0202359. doi: 10.1371/journal.pone.0202359. eCollection 2018. PMID 30183734